CLINICAL TRIAL: NCT06664905
Title: Impact of Different Resistance Training Protocols on Pain in Knee Osteoarthritis
Brief Title: Resistance Exercise in Severe Knee Osteoarthritis
Acronym: RTOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, José Casaña Granell, Head of the Physiotherapy Department, University of Valencia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OA-2023
Record Dates: First submitted 2023-04-14; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Knee Osteoarthritis
Keywords: Resistance Training; Knee Osteoarthritis; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Active Comparator): control, with no exercise
  Interventions: Other: Placebo
- 4 sets (Experimental): 4 sets of 10RM of knee extensions
  Interventions: Other: Resistance Exercise
- 8 sets (Experimental): 8 sets of 10RM of knee extensions
  Interventions: Other: Resistance Exercise
- 12 sets (Experimental): 12 sets of 10RM of knee extensions
  Interventions: Other: Resistance Exercise

INTERVENTIONS:
Other: Resistance Exercise — 10 Repetition Maximum (RM)
  Arms: 12 sets; 4 sets; 8 sets
Other: Placebo — No exercise
  Other Names: Control
  Arms: Placebo

SUMMARY:
This study aim to evaluate pain after different resistance training protocols (placebo, 4 sets of 10RM, 8 sets of 10 RM and 12 sets of 10RM) in patients with severe knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* men and women at least 55 years old
* diagnosed with severe knee OA
* scheduled for unilateral Total Knee Arthroplasty (TKA) surgery

Exclusion Criteria:

* pain in the contralateral (non-studied) limb (maximum ≥80 of 100 mm on a visual analog scale (VAS) during daily activities)
* another hip or knee joint replacement in the previous year
* any medical condition in which exercise was contraindicated
* participated in exercise programs (>2 days/week, training at intensities of 10-15RM) in the 6 months prior to the study
* history of stroke, brain surgery, major depression, or any self-perceived cognitive alterations that could affect the performance of study tasks

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Change in self-reported pain intensity | Pre-exercise (pre), immediate post exercise (post), and 10 min after exercise (post 10min)
  Measure of knee pain intensity with the Visual Analogue Scale (0-100mm), with higher scores reflecting higher perceived pain intensity
Change in pressure pain thresholds | Pre-exercise (pre), immediate post exercise (post), and 10 min after exercise (post 10min)
  Measured with a mechanical algometer (Wagner Instruments, Greenwich, CT, USA) in three sites (vastus medialis of the affected limb, vastus medialis of the unaffected limb, and distal to the non-dominant arm lateral epicondyle)

SECONDARY OUTCOMES:
WOMAC questionaire | pre-exercise
  A self-administered questionnaire for patients with hip or knee osteoarthritis. contain 24 items grouped into three dimensions: pain (5 items), stiffness (2 items) and physical function (17 items). Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Tampa Scale of Kinesiophobia (TSK 11) | pre-exercise
  Measure fear of movement and its score ranges from 11-44 with higher scores indicate an increasing degree of kinesiophobia
Chronic Pain Self-Efficacy Scale | pre-exercise
  Measures three domains of pain self-efficacy: pain management, physical functioning, and coping with symptoms management, physical functioning, and coping with symptomsmanagement, physical functioning, and coping with symptoms. A higher score suggests higher self-efficacy
Pain Catastrophizing Scale | pre-exercise
  People are asked to indicate the degree to which they have certain thoughts and feelings when they are experiencing pain using the 0 (not at all) to 4 (all the time) scale. A total score is yielded (ranging from 0-52), along with three subscale scores assessing rumination, magnification and helplessness, with higher scores reflecting worse condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic Universitary Hospital of Valencia, Valencia, Spain